CLINICAL TRIAL: NCT01524679
Title: A Prospective, Randomised, Open-label Phase IIb Clinical Trial Assessing the Effect of Pegylated Interferon Alfa-2a (Pegasys®)180 μg Once Weekly for 48 Weeks in Addition to an Ongoing Nucelos(t)Ide Based Treatment on Quantitative HBsAg Levels in Patients With Chronic HBeAg-negative Hepatitis B
Brief Title: Peg-interferon ADDed to an Ongoing Nucleos(t)Ide Based Treatment in Patients With Chronic Hepatitis B to Induce Decrease of HBs-Antigen
Acronym: PADD-ON
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Principal Investigator, Peter R. Galle, Univ.-Prof. Dr. med., Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML 27787
Record Dates: First submitted 2012-01-31; First posted 2012-02-02 (Estimated); Results first posted 2020-02-18 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Chronic Hepatitis B
Keywords: chronic hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment group (Experimental): pegylated interferon alfa-2a (Pegasys®) 180 μg once weekly for 48 weeks added to an ongoing nucleos(t)ide based treatment in patients with chronic HBeAg-negative hepatitis B
  Interventions: Drug: Pegylated interferon alfa-2a plus nucleos(t)ide(s)
- Control group (No Intervention): ongoing nucleos(t)ide based treatment alone

INTERVENTIONS:
Drug: Pegylated interferon alfa-2a plus nucleos(t)ide(s) — Pegylated interferon alfa-2a, s.c. 180 μg 1x/wk in addition to nucleos(t)ide(s)
  Other Names: Pegasys®
  Arms: Treatment group

SUMMARY:
A prospective, randomised, open-label phase IIb clinical trial assessing the effect of pegylated interferon alfa-2a(Pegasys®) 180 μg once weekly for 48 weeks added to an ongoing nucleos(t)ide based treatment in patients with chronic HBeAg-negative hepatitis B

The primary objective of the trial is to investigate whether the add-on of pegylated interferon alfa-2a to a continued treatment with nucleos(t)ide analogues increases the percentage of patients who have significant decrease (≥ 1log10) of HBs antigen after 48 weeks.

170 Patients with chronic hepatitis B, HBe antigen negative, already being treated with an oral antiviral regimen and having a nondetectable viral load for at least 12 months are included.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis B, HBe antigen negative
* treatment with a stable oral antiviral treatment (not containing telbivudine) and a fully suppressed viral load for at least 12 months (below limit of detection in conventional HBV-PCR assays, i.e. <116 IU / ml).
* 18-70 ys
* willingness and ability to give informed consent and to follow study procedures
* willingness to use adequate contraception

Exclusion Criteria:

* contraindications against treatment with pegylated interferon, e.g. depression, uncontrolled epilepsy, autoimmune diseases, pregnancy, leukocytopenia or thrombocytopenia at screening, etc.
* active alcohol or drug abuse
* preexisting polyneuropathy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2012-08; Primary Completion 2017-08-28 (Actual); Study Completion 2017-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter R. Galle, Univ.-Prof. Dr. med., Principal Investigator — I. Medizinische Klinik und Poliklinik, Universitätsmedizin Mainz
Locations (24):
- Germany (24):
  - Facharztpraxis Prof. Löhr, Wiesbaden, Hesse
  - Universitätsklinikum Aachen, Medizinische Klinik III, Aachen
  - Leber- und Studienzentrum am Checkpoint, Berlin
  - Charité Campus Virchow Klinikum, Universitätsmedizin Berlin, Berlin
  - Medizinische Klinik und Poliklinik I, Universitätsklinik Bonn, Bonn
  - Klinik für Gastroenterologie und Hepatologie am Abdominalzentrum Universitätsklinikum Köln, Cologne
  - Medizinisches Versorgungszentrum Dr. Mauss, Schmutz, Dr. Athmann, Dr. Hegener, Düsseldorf
  - Medizinische Klinik I, Klinik der J.W. Goethe Universität, Frankfurt
  - Teuber Consulting & Research KG, Frankfurt
  - Universitätsklinikum Freiburg Innere Medizin II, Freiburg im Breisgau
  - Universitätsklinikum Gießen und Marburg GmbH, Giessen
  - Universitätsklinikum Hamburg-Eppendorf, I. Med. Klinik und Poliklinik, Hamburg
  - Medizinische Hochschule Hannover, Klinik für Gastroenterologie, Hepatologie und Endokrinologie, Hanover
  - Universitätsklinikum Heidelberg, Medizinische Klinik IV, Heidelberg
  - Universitätsklinikum des Saarlandes, Homburg
  - Universitätsklinik Schleswig-Holstein Campus Kiel Klinik für Allgemeine Innere Medizin, Kiel
  - Universitätsklinikum Leipzig AöR, Leipzig
  - Universitätsmedizin Mainz, I. Med. Klinik und Poliklinik, Mainz
  - Universitätsklinikum Mannheim, Mannheim
  - Klinikum rechts der Isar der Technischen Universität München, München
  - Universitätsklinikum Regensburg, Regensburg
  - Uniklinik Tübingen Innere Medizin Abt. I, Tübingen
  - Universitätsklinikum Ulm, Zentrum für Innere Medizin, Ulm
  - Klinikum der Universität Würzburg Zentrum für Innere Medizin (ZIM) Medizinische Klinik und Poliklinik II Leber- und Infektionsambulanz, Würzburg

REFERENCES:
- [Background] Sprinzl MF, Grambihler A, Kittner JM, Wachtlin D, Ruckes C, et al. (2015) Prospective Randomized Open-label Trial Protocol Investigating the Addition of Pegylated Interferon-alpha to an Ongoing Nucleos(t)ide Treatment Regimen of HBeAg Negative Chronic Hepatitis B Patients (PADD-ON). J Clin Trials 5: 226. doi:10.4172/2167-0870.1000226

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Group | Control Group
Started | 112 | 58
Completed | 89 | 49
Not Completed | 23 | 9
Not completed — Lost to Follow-up | 1 | 4
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Adverse Event | 9 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Lack of Efficacy | 2 | 0
Not completed — e.g.wish for children, relocation | 6 | 1

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population is the modified ITT population consisting of all randomized patients with at least one available post-baseline assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Control Group | Total
Number analyzed (Participants) | 110 | 55 | 165
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (9.6) | 45.1 (9.7) | 44.3 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 16 | 42
  Male | 84 | 39 | 123
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 15 | 6 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 6 | 13
  White | 85 | 39 | 124
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  Germany | 110 | 55 | 165
Virology: HBV DNA quant. negative? [Count of Participants; unit: Participants]
  Yes | 109 | 54 | 163
  No | 1 | 1 | 2
Virology: Anti-HBs [Count of Participants; unit: Participants]
  Positive | 7 | 2 | 9
  Negative | 103 | 53 | 156
Virology: HBeAg [Count of Participants; unit: Participants]
  Positive | 0 | 0 | 0
  Negative | 110 | 55 | 165
Virology: Anti-HBe [Count of Participants; unit: Participants] — Population: Measure was not determined by the laboratory in 3 cases.
  Participants
    number analyzed (Participants) | 107 | 55 | 162
    Positive | 96 | 45 | 141
    Negative | 11 | 10 | 21
Virology: Anti-HBc [Count of Participants; unit: Participants] — Population: Measure was not determined by the laboratory in one case.
  Participants
    number analyzed (Participants) | 109 | 55 | 164
    Positive | 94 | 48 | 142
    Negative | 15 | 7 | 22
Virology: HCV [Count of Participants; unit: Participants]
  Positive | 0 | 0 | 0
  Negative | 110 | 55 | 165
Virology: HDV [Count of Participants; unit: Participants]
  Positive | 0 | 0 | 0
  Negative | 110 | 55 | 165
Virology: HIV [Count of Participants; unit: Participants] — Population: Measure was not determined by the laboratory in one case.
  Participants
    number analyzed (Participants) | 109 | 55 | 164
    Positive | 0 | 0 | 0
    Negative | 109 | 55 | 164
HBV Genotype known? [Count of Participants; unit: Participants]
  Yes | 22 | 12 | 34
  No | 88 | 43 | 131
HBV Genotype [Count of Participants; unit: Participants] — Population: The Genotype was only available in 34 patients.
  Participants
    number analyzed (Participants) | 22 | 12 | 34
    Genotype A | 2 | 1 | 3
    Genotype C | 1 | 0 | 1
    Genotype D | 16 | 11 | 27
    Genotype E | 1 | 0 | 1
    Wildtype | 1 | 0 | 1
    Not specified | 1 | 0 | 1
HBsAG Concentration [Mean (Standard Deviation); unit: IU/mL] — Population: HBsAG was not determined by the laboratory in 4 patients.
  IU/mL
    number analyzed (Participants) | 107 | 54 | 161
    (all) | 6547.5 (10326.2) | 8434.9 (12660.1) | 7180.6 (11159.5)

OUTCOME MEASURES:

1. Primary Outcome: Difference in Percentage of Patients Between Treatment and Comparator Arm Reaching a ≥ 1log10 Decline of Quantitative HBsAg After 48 Weeks
Description: Difference in percentage of patients between treatment and comparator arm reaching a ≥ 1log10 decline (tenfold reduction) of quantitative HBsAg after 48 weeks
Time Frame: 48 weeks
Population: mITT population consisting of all randomized patients with at least one post-baseline measurement
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 106 | 54
Participants
  Yes | 26 | 1
  Missing | 80 | 53
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; Nullhypothesis was the equality of response rates of the treatment group and the control group. Treatments were compared by a two-sided Fisher test on a level of significance of 0.05. The study was appropriately powered (80%) for this analysis; Test type: Superiority — The Fisher Test with asymptotic test statistic provided by the analysis software was used; p < 0.0001, Fisher Exact — This was the only a priori defined primary endpoint. There was no adjustment for multiple comparisons; There was no adjustment for other variables intended for the primary analysis. Confounding variables were analysed in subsequent analyses

2. Secondary Outcome: Change in Quantitative HBs Antigen at Week 12
Description: Change in quantitative HBs antigen at week 12. The data were log transformed before analysis and the changes to baseline were analysed. Therefore, the reported values might be interpreted as percentage changes. Lower scores mean a better outcome.
Time Frame: week 12
Population: Values were only available in 154 patients.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: IU/ml
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 101 | 53
IU/ml | 0.7058 [0.5803 to 0.8585] | 0.9380 [0.7154 to 1.2297]
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; Test type: Superiority; p = 0.0957, ANCOVA; Mean Difference (Final Values) = 0.7525, 95% CI 2-sided [0.5382 to 1.0521]

3. Secondary Outcome: Change in Quantitative HBs Antigen at Week 24
Description: Change in quantitative HBs antigen at week 24. The data were log transformed before analysis and the changes to baseline were analysed. Therefore, the reported values might be interpreted as percentage changes. Lower scores mean a better outcome.
Time Frame: week 24
Population: Values were only available in 151 patients.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: IU/ml
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 99 | 52
IU/ml | 0.3694 [0.2872 to 0.4752] | 0.7995 [0.5646 to 1.1322]
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; Test type: Superiority; p = 0.0005, ANCOVA; Mean Difference (Final Values) = 0.4621, 95% CI 2-sided [0.4621 to 0.7106]

ADVERSE EVENTS:
Time Frame: 48 weeks
Arm/Group | Treatment Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/112 | 0/58
Serious Adverse Events (participants affected / at risk) | 13/112 | 4/58
Other Adverse Events (participants affected / at risk) | 106/112 | 20/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=112) | Control Group (N=58)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
retinal haemorrhage (Eye disorders) | 1 (1) | 0 (0)
internal fixation of fracture (Surgical and medical procedures) | 1 (1) | 0 (0)
coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
chlamydial infection (Infections and infestations) | 1 (1) | 0 (0)
hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
hepatocellular lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
pain (General disorders) | 1 (1) | 0 (0)
pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
nasal tubinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=112) | Control Group (N=58)
chills (General disorders) | 11 (19) | 0 (0)
fatigue (General disorders) | 48 (52) | 2 (2)
influenza like illness (General disorders) | 13 (21) | 2 (2)
injection site erythema (General disorders) | 11 (12) | 0 (0)
pyrexia (General disorders) | 25 (28) | 0 (0)
arthralgia (Musculoskeletal and connective tissue disorders) | 31 (45) | 0 (0)
back pain (Musculoskeletal and connective tissue disorders) | 15 (17) | 2 (3)
myalgia (Musculoskeletal and connective tissue disorders) | 19 (21) | 0 (0)
nasopharyngitis (Infections and infestations) | 28 (31) | 3 (3)
abdominal pain upper (Gastrointestinal disorders) | 11 (11) | 6 (10)
diarrhoea (Gastrointestinal disorders) | 9 (12) | 1 (1)
nausea (Gastrointestinal disorders) | 12 (13) | 1 (1)
dizziness (Nervous system disorders) | 11 (18) | 0 (0)
headache (Nervous system disorders) | 40 (48) | 0 (0)
alopecia (Skin and subcutaneous tissue disorders) | 17 (17) | 0 (0)
dry skin (Skin and subcutaneous tissue disorders) | 7 (7) | 0 (0)
pruritus (Skin and subcutaneous tissue disorders) | 15 (17) | 0 (0)
rash (Skin and subcutaneous tissue disorders) | 8 (10) | 0 (0)
insomnia (Psychiatric disorders) | 9 (10) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 2 (2)
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 0 (0)
transaminases increased (Investigations) | 6 (9) | 0 (0)
weight decreased (Investigations) | 8 (8) | 1 (1)
thrombocytopenia (Blood and lymphatic system disorders) | 8 (11) | 0 (0)
decreased appetite (Metabolism and nutrition disorders) | 6 (9) | 0 (0)
erectile dysfunction (Reproductive system and breast disorders) | 6 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2013-04-19): https://cdn.clinicaltrials.gov/large-docs/79/NCT01524679/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-22): https://cdn.clinicaltrials.gov/large-docs/79/NCT01524679/SAP_001.pdf